CLINICAL TRIAL: NCT05975424
Title: A Long-term Follow-up Study of Subjects With Cervical Spinal Cord Injuries Who Received AST-OPC1 in Protocol AST-OPC1-01
Brief Title: LTFU Study of Subjects With Cervical SCI Who Received AST-OPC1
Status: Active, not recruiting | Type: Observational
Sponsor: Lineage Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AST-OPC1-02
Record Dates: First submitted 2023-05-24; First posted 2023-08-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for immune response monitoring and xenotransplantation safety samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects treated with AST-OPC1 in the initial dosing study AST-OPC1-01: Subjects treated with AST-OPC1 in the initial dosing study AST-OPC1-01 will be followed for 15-year long-term safety monitoring
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Observational study; annual MRI for first 5 years only to monitor changes in the injection site

SUMMARY:
This is a LTFU study for cervical SCI subjects that were administered AST-OPC1 cells in the main study AST-OPC1-01.

DETAILED DESCRIPTION:
Study AST-OPC1-02 is a Phase 1/2a open-label, multi-center long term follow-up (LTFU) study for twenty-five (25) subjects with cervical SCI that were administered AST-OPC1 cells in the main dose-escalation study AST-OPC1-01. The purpose of this study is to monitor long-term safety in subjects for 15 years post AST-OPC1 administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received AST-OPC1 under Study AST-OPC1-01
* Reconfirmation of consent for long-term follow-up

Exclusion Criteria:

•Subjects who, for geographic or compliance reasons, are inappropriate candidates for participation in a long-term follow-up study in the opinion of the Investigator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received administration of AST-OPC1 under clinical study protocol AST-OPC1-01
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2033-01-14 (Estimated); Study Completion 2033-01-14 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 15 years after AST-OPC1 injection
  Information will be collected on all adverse events through Year 5 and on late-occurring adverse events (Years 6-15) related to any changes in neurological condition, a fever of unknown etiology, and the development of neoplasias and/or neurological disorders.
Changes from baseline greater than 1.5x or 2x in chemistry and hematology panel results over 5 years after injection of AST-OPC1 | Up to 5 years after AST-OPC1 injection
  Summary statistics will be tabulated for chemistry and hematology laboratory parameter results and change from baseline to Year 5, as applicable, by cohort and overall. A table counting abnormal flags based on the respective lab's reference ranges by time point will be generated for each cohort and overall. At each visit, for each parameter, the number of subjects with low, normal, high, and clinically significant assessments will be tabulated.
Changes at the injection site as monitored by MRI | Up to 5 years after AST-OPC1 injection
  MRI scans will monitor the brain and cervical spine for any possible long-term changes that could be related to AST-OPC1

SECONDARY OUTCOMES:
Changes in neurologic function as assessed by the ISNCSCI | Up to 5 years after AST-OPC1 injection
  Subject baseline results will be compared against changes in motor and sensory examination results

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hogge, DVM, MS, PhD, Study Chair — Lineage Cell Therapeutics, Inc.
Locations (6):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Shepherd Center, Atlanta, Georgia
  - RUSH University Medical Center, Chicago, Illinois
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fessler RG, Ehsanian R, Liu CY, Steinberg GK, Jones L, Lebkowski JS, Wirth ED, McKenna SL. A phase 1/2a dose-escalation study of oligodendrocyte progenitor cells in individuals with subacute cervical spinal cord injury. J Neurosurg Spine. 2022 Jul 8;37(6):812-820. doi: 10.3171/2022.5.SPINE22167. Print 2022 Dec 1. PMID 35901693
- See also: A phase 1/2a dose-escalation study of oligodendrocyte progenitor cells in individuals with subacute cervical spinal cord injury — https://pubmed.ncbi.nlm.nih.gov/35901693/